CLINICAL TRIAL: NCT06497127
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of Subcutaneously Administered BW-00112 in Patients With Mixed Dyslipidemia
Brief Title: A Study in Patients With Mixed Dyslipidemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Argo Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BW-00112-2002
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): BW-00112 150 mg or volume-matched placebo on Day 1 and Day 90
  Interventions: Drug: BW-00112
- Cohort 2 (Experimental): BW-00112 300 mg or volume-matched placebo on Day 1 and Day 90
  Interventions: Drug: BW-00112
- Cohort 3 (Experimental): BW-00112 600 mg or volume-matched placebo on Day 1 and Day 90
  Interventions: Drug: BW-00112

INTERVENTIONS:
Drug: BW-00112 — BW-00112 or volume-matched placebo on Day 1 and Day 90

SUMMARY:
A Phase 2 in Patients With Mixed Dyslipidemia

DETAILED DESCRIPTION:
A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of Subcutaneously Administered BW-00112 in Patients with Mixed Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent and be able to comply with all study requirements.
2. Males or females aged 18 to 75 aged years, inclusive, at the time of informed consent
3. Fasting LDL-C ≥ 70 mg/dL [1.8 mmol/L] at Screening.

4.150 mg/dL [1.7 mmol/L] ≤ fasting TG < 500 mg/dL [5.6 mmol/L] at Screening, which may be repeated once if deemed necessary.

5.On a stable statin for at least 1 month before Screening and plan to remain on the same medication and dose for the duration of the study.

6.Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal 7.Male patients agreeing to use acceptable methods of contraception

Exclusion Criteria:

1. Active pancreatitis within 12 weeks prior to Day 1.
2. Clinically significant acute cardiovascular even or procedure
3. HbA1c > 9.0% at Screening or patients with diabetes who have experienced diabetic ketoacidosis, diabetic decompensation, hyperosmolar hyperglycemic nonketotic coma, diabetes complications, recurrent infections, or hospitalization related to poor glycemic control within 24 weeks prior to Day 1.
4. Presence of any clinically significant uncontrolled disease known to influence serum lipids or lipoproteins. NOTE: Patients on thyroid replacement therapy are eligible if the dosage of thyroxine has been stable for at least 12 weeks prior to Day 1.
5. Use of TG lowering medication , non-prescription dietary supplements or other cholesterol lowering medication 30 days prior to Day 1, other than statins and ezetimibe.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in fasting TG | From baseline to Day 180
  Percent change in fasting TG from baseline to Day 180

SECONDARY OUTCOMES:
Percent change in fasting TG | From baseline to Day 15, 30, 60, 90, 135, 225, and 270
  Percent change in fasting TG from baseline to Day 15, 30, 60, 90, 135, 225, and 270

CONTACTS AND LOCATIONS:
Overall Officials: Yuqiong Li, Master, Study Director — Shanghai Argo Biopharmaceutical Co., Ltd.
Locations (14):
- United States (14):
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Excel Medical Clinical Trials, LLC, dba Flourish Research, Boca Raton, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Clinical Site Partners Leesburg, LLC dba Flourish Research, Leesburg, Florida
  - Suncoast Research Group, LLC DBA Flourish Research, Miami, Florida
  - Clinical Site Partners, LLC DBA Flourish Research, Miami, Florida
  - East Coast Institute for Research LLC, Canton, Georgia
  - Alliance for Multispecialty Research, LLC, Oak Brook, Illinois
  - Alliance for Multispecialty Research, LLC, Park Ridge, Illinois
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No